CLINICAL TRIAL: NCT01289912
Title: Randomized Double-Blind Phase 2 Trial Of RAD001 For Neurocognition In Individuals With Tuberous Sclerosis Complex
Brief Title: Trial of RAD001 and Neurocognition in Tuberous Sclerosis Complex (TSC)
Acronym: TSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mustafa Sahin (Other)
Collaborators: Tuberous Sclerosis Alliance (Other); Autism Speaks (Other); Novartis Pharmaceuticals (Industry); Seizure Tracker LLC (Unknown)
Responsible Party: Sponsor-Investigator, Mustafa Sahin, MD, PhD, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-06-0247
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex; Autism; Neurocognition; RAD001; Everolimus; Afinitor; TSC
MeSH Terms: conditions — Tuberous Sclerosis; Autistic Disorder | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAD001 (Experimental): RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  Interventions: Drug: RAD001
- Placebo (Placebo Comparator): Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAD001 — RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
  Other Names: Everolimus; Afinitor
  Arms: RAD001
Drug: Placebo — Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
  Arms: Placebo

SUMMARY:
Tuberous Sclerosis Complex (TSC) is a multi-system disease, usually presenting with seizures, mental retardation and autism, and exhibiting a high variability in clinical findings both among and within families. Investigators are doing research in order to identify possible neurocognitive benefits from treatment with RAD001 or placebo for a six month period. There may also be potential for improvements in seizure frequency, sleep and autistic behaviors. We hope this trial will lead to a better understanding of TSC and to new forms of treatment, to benefit children and adults with TSC in the future.

Individuals diagnosed with TSC will be asked to participate in this study if they are between the ages of 6 and 21 years of age and have an IQ of greater than or equal to 60. Both males and females will be asked to participate. Additionally, to be eligible for study participation, individuals must have been on the same seizure medication(s), if applicable, for at least 6 months. Individuals must also be able to participate in neuropsychological testing and meet certain medical criteria. They will need to sign an informed consent. If enrolled in the study, participants will have a number of screening tests to help determine if they are eligible for participation in the clinical trial. If eligible for the treatment phase of the trial, they will be asked to take either the study drug or a placebo (pill with no medicine), which is determined by chance.

The study involves about 9 visits, 3 of which can be done locally, over a six month period, as well as follow-up calls with our research nurse. Study visits will vary in length. Screening, three month and six month visits may last up to 8 hours, while all other visits will be less than 2 hours. The study visits include blood draws, laboratory tests and neuropsychological assessments. There is no fee to participate in this study. The study drug will be provided at no charge during the study.

After all study data has been analyzed, families will be informed of the overall results. Treatment on this study may or may not improve a child's learning skills (neurocognition). Future patients may benefit from what is learned.

DETAILED DESCRIPTION:
This is a signal-seeking Phase II randomized, placebo-controlled trial of RAD001 in children and young adults with TSC with neurocognition as the primary outcome and autism spectrum disorder as a secondary outcome.

Specific Aims /Objectives Primary objective

* To evaluate the efficacy of RAD001 on neurocognition in patients with TSC compared to placebo as measured by well-validated, standardized, direct and indirect neurocognitive tools.
* To evaluate the safety of RAD001 compared with placebo in patients with TSC focusing on NCI CTCAE Grade 3 and 4 adverse events, serious adverse events, and Grade 3 and 4 laboratory toxicities.

Secondary objectives

* Comparison of absolute change from baseline in frequency of epileptiform events as recorded on seizure diaries between patients taking RAD001 vs. placebo
* Comparison of sleep disturbances between patients taking RAD001 vs. placebo, measured by the Pediatric Sleep Questionnaire (PSQ) and sleep logs
* Comparison of autism spectrum disorders features between patients taking RAD001 vs. placebo, measured by ADOS and SRS
* Comparison of academic skills between patients taking RAD001 vs. placebo, measured by WRAT4
* Comparison of behavioral problems between patients taking RAD001 vs placebo, measured by behavioral rating scales (BRIEF, BASC, SDQ, CHQ and SRS)

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients ages 6 to 21 years of age.
2. IQ ≥60.
3. Ability to participate in direct neuropsychological and developmental testing.
4. English as primary language.
5. Diagnosis of tuberous sclerosis complex confirmed by genetic testing and/or clinically definite diagnosis of tuberous sclerosis complex according to the modified Gomez criteria and an IQ>60.
6. Stable anti-epileptic drugs (no changes in medications except dose for >6 months).
7. Adequate renal function. The GFR would be greater than 50 ml/min.m2 as determined by the Schwartz Formula for children and MDRD for adults:

   http://www.nkdep.nih.gov/professionals/gfr_calculators/index.htm
8. If female and of child bearing potential, documentation of negative pregnancy test prior to enrollment. Sexually active pre-menopausal female patients (and female partners of male patients) must use adequate contraceptive measures, excluding estrogen containing contraceptives, while on study. Abstinence will be considered an adequate contraceptive measure.
9. INR ≤1.5 (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for >2 weeks at time of randomization.)
10. Adequate liver function as shown by:

    * serum bilirubin ≤ 1.5 x ULN
    * ALT and AST ≤ 2.5x ULN (≤ 5x ULN in patients with liver metastases)
11. Written informed consent according to local guidelines.

Exclusion criteria:

1. Change of one or more antiepileptic medication in the past 6 months.
2. Prior exposure to the systemic use of an mTOR inhibitor.
3. Exposure to any investigational agent in the 30 days prior to randomization.
4. Neurosurgery within 6 months.
5. Known impaired lung function (e.g.FEV1 or DLCO <70% of predicted), if not resolved or if resolved within past 24 months.
6. Significant hematological or hepatic abnormality (i.e. transaminase levels > 2.5 x ULN or serum bilirubin > 1.5 x ULN, hemoglobin < 9 g/dL, platelets < 80,000/ mm3, absolute neutrophil count < 1,000/mm3).
7. Serum creatinine > 1.5 x ULN.
8. Uncontrolled hyperlipidemia: Fasting serum cholesterol > 300 mg/dL OR > 7.75 mmol/L AND Fasting triglycerides > 2.5 x ULN.
9. Uncontrolled diabetes mellitus as defined by fasting serum glucose > 1.5 x ULN.
10. Patients with bleeding diathesis or on oral anti-vitamin K medication (except low dose warfarin).
11. Patients with known history of HIV seropositivity.
12. Pregnancy or breast feeding.
13. Active infection at date of randomization.
14. Prior history of organ transplant.
15. Recent surgery (involving entry into a body cavity or requiring sutures) within the 4 weeks prior to randomization.
16. Inability to attend scheduled clinic visits.
17. History of malignancy in the past two years, other than squamous or basal cell skin cancer.
18. Patients should not receive immunization with attenuated live vaccines within one month of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
19. Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).

    Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV DNA and HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.
20. Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
21. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * symptomatic congestive heart failure of New York heart Association Class III or IV
    * unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
22. Patients who have received an IQ score under 60 in the six months prior to the study screening visit will be deemed ineligible.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Sahin, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- See also: Tuberous Sclerosis Alliance — http://www.tsalliance.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
- Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time (delete: each day) in the morning after a light, nonfat breakfast.
Period: Overall Study
Arm/Group | RAD001 | Placebo
Started | 32 | 15
Completed | 29 | 13
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RAD001 | Placebo | Total
Number analyzed (Participants) | 32 | 15 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.25 (5.06) | 11.47 (5.30) | 12.68 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 23
  Male | 16 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Safety of RAD001 on Neurocognition in Patients With TSC Compared With Placebo in Patients With TSC.
Description: Evaluation of the safety of RAD001 compared with placebo in patients with TSC focusing on NCI CTCAE Grade 3 and 4 adverse events, serious adverse events, and Grade 3 and 4 laboratory toxicities.
Time Frame: 6 months
Measure: Number; unit: Adverse Events
Arm/Group | RAD001 | Placebo
Number analyzed (Participants) | 32 | 15
Adverse Events | 325 | 147

2. Primary Outcome: Evaluation of the Efficacy of RAD001 on Neurocognition in Patients With TSC Compared With Placebo.
Description: Baseline and 6 month Timepoint scores are reported for the following primary outcome measures:
  1. Peabody Picture Vocabulary Test 4 (PPVT-4; Receptive Language Measure). Scores reported as (mean, SD). Range=40-160, higher scores are better.
  2. Expressive Vocabulary Test 2 (EVT-2; Expressive Language Measure). Scores reported as (mean, SD). Range=40-160, higher scores are better.
  3. Wide Range Assessment of Memory and Learning 2 (WRAML2; Measure of Verbal Memory and Attention ). Scores reported as (mean, SD). Range=1-19, higher scores are better.
  4. Vineland Adaptive Behavior Scales-II (VABS-II; Measure of Adaptive Behavior). Scores reported as (mean, SD). Range = 40-160, higher scores are better.
  5. Purdue Pegboard Test (Measure of Fine Motor Speed and Coordination). Scores reported as (mean, SD). Range = 40-160, higher scores are better.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo - Baseline: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
- RAD001 - Baseline: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
- Placebo - 6 Months: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- RAD001 - 6 Months: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
Arm/Group | Placebo - Baseline | RAD001 - Baseline | Placebo - 6 Months | RAD001 - 6 Months
Number analyzed (Participants) | 15 | 32 | 13 | 29
units on a scale
  PPVT4 (Receptive Language) | 86.00 (17.78) | 81.06 (23.96) | 88.54 (17.21) | 82.5 (22.32)
  EVT2 (Expressive Language) | 85.47 (12.22) | 90.00 (21.15) | 89.15 (16.08) | 82.55 (21.22)
  WRAML2 Verbal Learning | 8.00 (2.00) | 7.14 (3.16) | 8.46 (2.44) | 7.85 (2.92)
  WRAML2 Verbal Recall | 7.07 (2.94) | 7.52 (2.53) | 8.23 (3.49) | 8.08 (2.77)
  VABS2 Adaptive Behavior Composite | 78.79 (19.69) | 72.06 (13.90) | 79.00 (15.26) | 74.72 (14.57)
  VABS2 Communication | 81.27 (21.87) | 73.68 (15.45) | 81.77 (16.66) | 76.79 (14.76)
  VABS2 Socialization | 79.07 (19.67) | 74.10 (15.46) | 80.38 (17.78) | 76.86 (16.40)
  VABS2 Daily Living Skills | 78.80 (19.50) | 74.68 (15.69) | 81.69 (14.74) | 76.41 (17.37)
  VABS2 Motor Skills | 89.87 (18.26) | 78.83 (21.68) | 92.69 (18.65) | 87.79 (18.12)
  Pegboard, Dominant Hand | 101.33 (54.27) | 103.06 (41.18) | 89.83 (24.99) | 97.25 (39.02)
  Pegboard, Non-Dominant Hand | 105.27 (37.10) | 119.30 (44.19) | 92.15 (34.26) | 112.78 (50.89)

3. Primary Outcome: Evaluation of the Efficacy of RAD001 on Neurocognition (Cambridge Neuropsychological Test Automated Battery) in Patients With TSC Compared With Placebo.
Description: Scores are reported for baseline and 6 month timepoints on the Cambridge Neuropsychological Test Automated Battery (CANTAB) subscales below. For all subscales, scores are reported as the mean difference between the study subjects and a normative population matched for age, gender and IQ (e.g., subject subscale score - mean of matched normative group = reported score). Higher scores represent a better outcome.
  1. Spatial Span (SSP) (spatial memory span) Range: -3 to 3
  2. Spatial Working Memory (working memory) Range: -3 to 3
  3. Pattern Recognition Memory (PRM) (visual pattern recognition memory) Range: -3 to 3
  4. Spatial Recognition Memory (SRM) (spatial recognition memory) Range: -4 to 4
  5. Rapid Visual Information Processing (RVIP) (sustained attention) Range: -4 to 4
  6. Stockings of Cambridge (SOC) (spatial planning) Range: -4 to 4
  7. Intra-Extra Dimensional Set Shift (IDED) (cognitive flexibility) Range: -5 to 5
  8. Reaction Time (processing speed) Range: -5 to 5
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo - Baseline: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Baseline.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
- RAD001 - Baseline: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. Baseline.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- Placebo - 6 Months: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. 6 months.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- RAD001 - 6 Months: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. 6 months.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
Arm/Group | Placebo - Baseline | RAD001 - Baseline | Placebo - 6 Months | RAD001 - 6 Months
Number analyzed (Participants) | 15 | 32 | 13 | 29
units on a scale
  CANTAB Pattern Recognition Memory | -1.48 (1.9) | -1.23 (2.11) | -.91 (1.6) | -1.09 (1.79)
  CANTAB Spatial Recognition Memory | -2.33 (1.4) | -2.24 (1.33) | -2.62 (1.58) | -2.19 (1.56)
  CANTAB Spatial Span | -1.32 (1.18) | -1.02 (1.20) | -1.29 (1.41) | -1.32 (1.37)
  CANTAB Spatial Working Memory | -.66 (.79) | -.67 (1.57) | -.73 (.97) | -.27 (2.87)
  CANTAB Reaction Time | -2.24 (3.63) | -1.15 (2.22) | -.88 (1.38) | -2.91 (3.84)
  CANTAB Rapid Visual Processing | -.96 (2.59) | -1.41 (2.8) | -.97 (2.71) | -1.2 (2.15)
  CANTAB Stockings of Cambridge | -1.38 (1.32) | -1.89 (1.47) | -.58 (1.11) | -1.84 (1.32)
  CANTAB IDED | -1.02 (1.65) | -1.48 (2.05) | -1.05 (1.64) | -2.24 (3.32)

4. Secondary Outcome: Comparison of Absolute Change From Baseline in Frequency of Epileptiform Events Between Patients Taking RAD001 vs. Placebo
Description: Comparison of absolute change from baseline in frequency of epileptiform events as recorded on seizure diaries between patients taking RAD001 vs. placebo
Time Frame: 6 months
Population: Data was not collected reliably and therefore was not analyzed.
Groups:
- RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis.
  RAD001: RAD001 is formulated as tablets of 5.0 mg strength, blister-packed under aluminum foil in units of 10 tablets and dosed on a regular basis. RAD001 tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of RAD001 orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
- Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10.
  Placebo: Matching placebo will be provided as a matching tablet and will also be blister packed under aluminum foil in units of 10. Matching placebo tablets should be opened only at the time of administration as drug is both hygroscopic and light-sensitive.
  Patients will be instructed to take 4.5 mg/m2 of the matching placebo orally with a glass of water at regular intervals at the same time in the morning after a light, nonfat breakfast.
Arm/Group | RAD001 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Comparison of Sleep Disturbances Between Patients Taking RAD001 vs. Placebo
Description: Comparison of sleep disturbances between patients taking RAD001 vs. placebo, measured by the Pediatric Sleep Questionnaire (PSQ) and sleep logs
Time Frame: 6 months
Population: Data was not collected reliably and therefore was not analyzed.
Arm/Group | RAD001 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Comparison of Autism Spectrum Disorders Features Between Patients Taking RAD001 vs. Placebo
Description: Scores for the Baseline and 6 Month Timepoints are reported. The secondary outcome measure was the Social Responsiveness Scale (SRS). Standard scores are reported with a mean of 100 and standard deviation of 15. The range is 40-160 with higher scores indicating a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale (SRS)
Arm/Group | Placebo - Baseline | RAD001 - Baseline | Placebo - 6 Months | RAD001 - 6 Months
Number analyzed (Participants) | 15 | 32 | 13 | 29
units on a scale (SRS)
  SRS Social Responsiveness (range 40(worse) -160) | 77.14 (17.50) | 76.43 (18.62) | 80.62 (22.83) | 75.69 (19.27)
  SRS Social Awareness | 67.40 (14.69) | 62.90 (15.32) | 67.38 (15.51) | 64.86 (17.19)
  SRS Social Cognition | 76.43 (19.59) | 75.70 (18.77) | 81.15 (18.86) | 76.17 (18.98)
  SRS Social Communication | 74.36 (16.75) | 72.23 (17.18) | 76.85 (21.55) | 71.69 (17.98)
  SRS Social Motivation | 69.80 (16.60) | 69.60 (14.76) | 72.77 (20.77) | 67.24 (16.37)
  SRS Autism Mannerisms | 76.71 (17.32) | 80.03 (20.24) | 79.77 (24.50) | 78.66 (20.16)

7. Secondary Outcome: Comparison of Academic Skills Between Patients Taking RAD001 vs. Placebo
Description: Scores are reported for Baseline and 6 Month Timepoints. The secondary outcome measure was the Wide Range Achievement Test 4 (WRAT4), which was used to assess academic skills. The Reading and Math subtests were used. Standard scores are reported which have a mean of 100 and a standard deviation of 15 (range=40-160 where higher is better).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo - Baseline | RAD001 - Baseline | Placebo - 6 Months | RAD001 - 6 Months
Number analyzed (Participants) | 15 | 32 | 13 | 29
units on a scale
  Word Reading (WRAT 4) | 86.80 (16.79) | 84.28 (20.07) | 91.15 (20.76) | 84.45 (20.45)
  Math Computation (WRAT 4) | 76.00 (15.64) | 74.60 (17.99) | 77.31 (16.93) | 73.81 (16.01)

8. Secondary Outcome: Comparison of Behavioral Problems Between Patients Taking RAD001 vs Placebo
Description: Scores for Baseline and 6 Month Timepoints are reported for the following secondary outcome measures:
  1. Behavior Rating Inventory of Executive Function (BRIEF) (Measure of executive functions) T-scores are reported, with a mean of 50 and a standard deviation of 10. The range is 30-100 with higher scores indicating a worse outcome.
  2. Behavioral Assessment System for Children (BASC) (Measure of emotional and behavioral problems) T-scores are reported (mean of 50, SD of 10). The range is 30-100 with higher scores indicating a worse outcome. Conversely, on the Adaptive Skills subscale of the BASC, lower scores indicate a poorer outcome.
  3. Strengths and Difficulties Questionnaire (SDQ). Includes questions related to emotional symptoms, conduct problems, inattention/hyperactivity, peer relationship problems and prosocial behavior. Responses to these items are summed to comprise a Total Difficulties Score, which ranges from 0-40, with lower scores indicating a better outcome
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo - Baseline | RAD001 - Baseline | Placebo - 6 Months | RAD001 - 6 Months
Number analyzed (Participants) | 15 | 32 | 13 | 29
units on a scale
  BRIEF Global Executive Composite | 70.50 (15.13) | 69.48 (12.98) | 62.25 (12.53) | 64.68 (10.88)
  BRIEF Behavioral Regulation Index | 70.93 (16.89) | 66.53 (14.50) | 60.83 (12.41) | 62.57 (12.00)
  BRIEF Metacognition Index | 68.07 (14.52) | 68.93 (12.12) | 61.83 (12.97) | 64.57 (10.65)
  BASC2 Behavioral Symptoms Index | 62.29 (12.61) | 58.97 (10.87) | 57.54 (10.02) | 55.41 (11.26)
  BASC2 Externalizing Problems | 57.36 (15.58) | 53.24 (9.85) | 52.62 (9.26) | 52.34 (8.59)
  BASC2 Internalizing Problems | 58.43 (18.34) | 51.55 (12.09) | 56.00 (19.37) | 51.45 (14.42)
  BASC2 Adaptive Skills | 38.79 (13.16) | 36.72 (10.22) | 42.08 (13.27) | 40.00 (12.02)
  SDQ Total Difficulties Scale | 16.00 (6.93) | 15.46 (5.61) | 14.42 (5.09) | 13.20 (5.90)

ADVERSE EVENTS:
Arm/Group | RAD001 | Placebo
Serious Adverse Events (participants affected / at risk) | 3/32 | 0/15
Other Adverse Events (participants affected / at risk) | 30/32 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=32) | Placebo (N=15)
Septicemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
high fever/pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Personality/Behavior (Social circumstances) | 1 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 (N=32) | Placebo (N=15)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (18) | 5 (8)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (2)
Stomach ache/pain/upset/irritation (Gastrointestinal disorders) | 8 (11) | 6 (8)
Stomach flu (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 4 (4)
stomach bug/virus/flu (Gastrointestinal disorders) | 2 (2) | 2 (2)
Bloody nose/nosebleed (General disorders) | 2 (6) | 1 (5)
Body pain/swelling/generalized pain NOS (General disorders) | 8 (8) | 3 (6)
Cavity (General disorders) | 0 (0) | 1 (1)
Cold (General disorders) | 8 (14) | 2 (3)
Cold Sores (General disorders) | 1 (1) | 1 (1)
Congestion (General disorders) | 1 (1) | 1 (5)
Cough (General disorders) | 7 (8) | 6 (11)
Fall (General disorders) | 1 (2) | 1 (1)
Fatigue (General disorders) | 7 (12) | 1 (2)
Feeling Cold (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 10 (17) | 4 (5)
Increased Energy (General disorders) | 0 (0) | 1 (1)
Ingrown toenail (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 3 (3) | 0 (0)
Muscle cramp/soreness (General disorders) | 2 (2) | 1 (2)
Runny nose (General disorders) | 4 (5) | 3 (4)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Ear Infection (Infections and infestations) | 3 (5) | 2 (2)
Mouth Sore (Infections and infestations) | 13 (28) | 5 (7)
Mouth Ulcer (Infections and infestations) | 8 (13) | 3 (5)
Mouth irritation/pain (Infections and infestations) | 4 (4) | 1 (3)
Painful Urination (Infections and infestations) | 0 (0) | 1 (1)
Sore throat (Infections and infestations) | 8 (9) | 2 (2)
Stomach Infection (Infections and infestations) | 2 (2) | 0 (0)
Strep throat (Infections and infestations) | 3 (4) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising/contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Cuts/Abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Soreness due to injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Loss of appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 13 (40) | 5 (18)
Seizures (Nervous system disorders) | 5 (7) | 1 (1)
Sleep Disturbance/Insomnia (Nervous system disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Behavioral/personality changes (Psychiatric disorders) | 5 (5) | 1 (1)
UTI/urinary frequency/incontinence (Renal and urinary disorders) | 7 (10) | 0 (0)
Genital irritation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Phlegm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stuffy nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection/Upper Airways NOS (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 3 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Abscess (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Acne/Pimples (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Athlete's foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Dry/itchy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash/hives (Skin and subcutaneous tissue disorders) | 10 (11) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Triglyceride-serum high (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No